CLINICAL TRIAL: NCT05751980
Title: Optimizing Medication Management by Older Adults Through the Med Wise Rx Community-based Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2022-1605; Pharmacy-Gen (Other: UW Madison); Protocol Version 1/9/2024 (Other: UW Madison); A561000 (Other: UW Madison)
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Communication Research
Keywords: Comprehensive Medication Review; Older Adults; Pharmacists; Multiple Medications

STUDY DESIGN:
Intervention Model Description: Wait-list control, a mixed-methods approach incorporating surveys, observational data collection, and interviews
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Med Wise Rx (Experimental): An evidence-informed two-session interactive behavioral workshop. Participants will begin intervention within 3 weeks of enrollment.
  Interventions: Behavioral: Med Wise Rx
- Waitlist Control (Active Comparator): Participants will be crossed over to Med Wise Rx intervention up to 2 months after enrollment.
  Interventions: Behavioral: Med Wise Rx

INTERVENTIONS:
Behavioral: Med Wise Rx — The program consists of two 120-minute classes led by trained community site-based facilitators, designed to help older adults communicate more effectively with their pharmacists.

SUMMARY:
This study's overall goal is to enhance older adults' communication skills to access medication information and services to manage their medications safely and effectively. Med Wise Rx is an online 2-session program to improve communication skills for accessing medication information and services, leading to improved medication management. 160 adults age 65 years or older taking 4 or more medications will be on study for up to 9 months.

DETAILED DESCRIPTION:
This study's overall goal is to enhance older adults' communication skills to access medication information and services to manage their medications safely and effectively. Older adults are 2-3 times more likely to experience adverse drug events (ADEs) which are linked to falls, morbidity, hospitalization, loss of independence and death. More complicated regimens, poor adherence and poor communication contribute to this greater risk.

The Med Wise Rx Program is an evidence-informed two-session interactive behavioral workshop that has been delivered in partnership with Aging and Disability Resource Centers (ADRCs) who informed the program design. This program was evaluated with 198 older adults in 8 Wisconsin counties and found a significant increase in participants' reported self-efficacy, communication skills and requests for medication checkups or comprehensive medication reviews (CMRs). There is a need for updating the Med Wise Rx program for dissemination virtually and to systematically examine the new design's effectiveness and implementation in organizations serving older adults.

The study team will conduct a Type 2 hybrid effectiveness-implementation study of Med Wise Rx delivered through a new technology-supported mode of education. A randomized patient to group treatment trial with a waitlist control group for older adults and/or caregivers aged 65 or older will be used. A mixed-methods approach will be used, incorporating surveys, observational data collection, and interviews. The RE-AIM Framework will guide and inform the processes. In collaboration with the Community Academic Aging Research Network (CAARN) and five community partners associated with 7 counties, this dissemination and implementation study will:

* AIM 1. Refine strategies to disseminate and implement the Med Wise Rx communication program through enhanced digital delivery methods.
* AIM 2. Develop a facilitator training program that maximizes Med Wise Rx delivery fidelity in its new format.
* AIM 3. Evaluate the reach, effectiveness, adoption/ acceptability, implementation/ enactment, and maintenance of the Med Wise Rx program delivery by Aging and Disability Resource Centers (ADRCs) and participants at 8 weeks and 6 months post-delivery.

Protocol Amendment 1/31/24 to remove 6-month follow up time point for cohorts enrolled this spring.

ELIGIBILITY:
Inclusion Criteria:

* community-dwelling
* age 65 or older
* use 4 or more medications
* must have the cognitive ability to participate
* speak and read English
* be able to use a computer

Exclusion Criteria:

* unable to attend either of the two Med Wise sessions (the first or the second, wait-listed control)
* under age 65
* unable to read/write English
* taking fewer than 4 chronic medications
* did not pass cognitive screener

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 121 (Actual)
Dates: Start 2023-01-23 (Actual); Primary Completion 2024-08-25 (Actual); Study Completion 2024-08-25 (Actual)

PRIMARY OUTCOMES:
Change in Number of Participant Reported CMRs | 8 weeks post-intervention (up to 12 weeks on study), 6 months post-intervention (up to 9 months on study for cohorts enrolled prior to Spring 2024)
  Specific questions included on survey tool will identify whether participant's report receiving a CMR, verifying (via protocol) Hometown Pharmacy CMRs reported.
Change in Communication Confidence measured by validated Participant Survey | baseline, 8 weeks post-intervention (up to 12 weeks on study), 6 months post-intervention (up to 9 months on study for cohorts enrolled prior to Spring 2024)
  The participant survey has 24 items and follows Bandura's self-efficacy theory and 0-10 scale. Total score (0-240) and individual items using repeated measures ANOVA will be used (survey administered at all 3 time points). Higher scores indicate increased communication confidence.
Change in Worries as measured by Participant Survey | baseline, 8 weeks post-intervention (up to 12 weeks on study), 6 months post-intervention (up to 9 months on study for cohorts enrolled prior to Spring 2024)
  The survey has 7-items scored on a 0-3 scale Total score of 0-21 with higher scores indicating increased worries.
Change in Knowledge about what a pharmacist can do to help as measured by Participant Survey | baseline, 8 weeks post-intervention (up to 12 weeks on study)
  Participant Survey has 6 items, scored yes, no, and unsure. A change in participant response for each item will be reported.
Change in Number of Services Requested | baseline, 8 weeks post-intervention (up to 12 weeks on study), 6 months post-intervention (up to 9 months on study for cohorts enrolled prior to Spring 2024)
  In addition to the participant CMR request, this measure captures the number of other reasons the participants have visited the pharmacist for.
Number of Changes in Medication List or Schedule | baseline, 8 weeks post-intervention (up to 12 weeks on study), 6 months post-intervention (up to 9 months on study for cohorts enrolled prior to Spring 2024)
  Changes in a medication list or schedule (i.e. time of day) that can improve medication safety and efficacy for older adults will be tallied.

CONTACTS AND LOCATIONS:
Overall Officials: Beth Martin, PhD, MS, RPh, FAPhA, Principal Investigator — University of Wisconsin, Madison
Locations (4):
- United States (4):
  - ADRC of Eau Claire County, Eau Claire, Wisconsin
  - Village of Greendale Public Health, Greendale, Wisconsin
  - Aging and Disability Resource Center (ADRC) of Kenosha County, Kenosha, Wisconsin
  - ADRC of Calumet, Outagamie & Waupaca County, Waupaca, Wisconsin

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2023-06-15): https://cdn.clinicaltrials.gov/large-docs/80/NCT05751980/ICF_000.pdf